CLINICAL TRIAL: NCT02538913
Title: Exercise Training for Rectal Cancer Patients. A Randomized Controlled Trial.
Brief Title: Exercise Training for Rectal Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too slow recruitment; lack of resources
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/2284
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Rectal Neoplasms
Keywords: Exercise; Pelvic floor; Prehabilitation; Fecal incontinence; Urinary incontinence; Sexual dysfunction, physiological
MeSH Terms: conditions — Rectal Neoplasms; Motor Activity; Fecal Incontinence; Urinary Incontinence; Sexual Dysfunction, Physiological | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Patients randomized to the exercise training group will be individually instructed in correct pelvic floor muscle contractions and intensive pelvic floor muscle training to perform daily. In addition they will be encouraged to exercise regularly ≥3 days/week. The exercise program will be individualized and consisting of both aerobic and strength exercise training.
  Interventions: Behavioral: Exercise training; Procedure: Usual care
- Usual care (Active Comparator): Patients randomized to the control group will receive standard care which does not include any pelvic floor muscle training or individualized exercise training
  Interventions: Procedure: Usual care

INTERVENTIONS:
Behavioral: Exercise training — Daily pelvic floor muscle training and individualized regular exercise training (aerobic and strength exercise) three days per week.
  Arms: Exercise training
Procedure: Usual care — Patients randomized to the control group will receive standard care which does not include any pelvic floor muscle training or individualized exercise training

SUMMARY:
Cancer treatments often cause acute toxicity during treatment, and late toxicity after treatments have ended. Bowel dysfunctions, incontinence (anal and urinary) and dysfunction are late side effects associated with cancer treatment in general, and patients treated for pelvic malignancies are at a higher risk. In Norway, the incidence of rectal cancer was 1329 in 2010. Advances in the treatment during the past few decades have led to fewer local recurrences and increased long-term survival, and today the relative survival is 66% for women and 64% for men. More patients are having sphincter-preserving surgery with low colorectal or ultralow coloanal anastomoses, and low anterior resection (LAR) is done in 70% of the patients with curative surgery. Unfortunately, many patients experience altered bowel function after LAR. Frequent bowel movements, urgency, evacuatory difficulties and fecal incontinence are common and distressing complications. These functional disturbances are seen in up to 50-60% of the patients, and most frequent when surgery is combined with neoadjuvant therapy. Urinary incontinence and decreased sexual function is also common in both men and women following rectal cancer treatment.

In many surgical settings, patients with higher preoperative physical fitness rehabilitate more quickly and have fewer operative complications compared with patients who are less physically fit. Additionally, specific strength training of the pelvic floor muscles builds up muscle volume, elevates the location of the pelvic floor muscles and pelvic organs, and closes the levator hiatus thus providing improved structural support for the pelvic floor as well as more optimal automatic function. The aim of the present trial is to investigate whether exercise training including pelvic floor muscle training during preoperative radiotherapy can reduce symptoms of bowel, urinary and sexual dysfunction and affect the physiology of the anal sphincter muscle after LAR. In addition quality of life, cardiopulmonary parameters and postoperative complications will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Cancer recti
* Planned curative LAR with preoperative radiotherapy
* Cancer stadium I-III
* Able to speak and understand Norwegian

Exclusion Criteria:

* Previous radiotherapy
* Previous pelvic surgery
* Diseases affecting the anal sphincter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Anal incontinence | 3 months post surgery
  St. Marks score

SECONDARY OUTCOMES:
Anal incontinence | 12 months post surgery
  St. Marks score
Urinary incontinence | 3 and 12 months post surgery
  International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI/SF)
Bowel dysfunction | 3 and 12 months post surgery
  Low anterior resection syndrome score (LARS)
Physiology of the anal sphincter | 3 and 12 months post surgery
  Anal manometry
Sexual dysfunction | 3 and 12 months post surgery
  The International Index of Erectile Function (IIEF) for men and the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire (PISQ-IR) (PISQ-IR) for women
Quality of life | 3 and 12 months post surgery
  The European Organization for Research and Treatment of Cancer Quality of Life core questionnaire (EORTC QLQ-C30) and the colorectal cancer specific Quality of Life Questionnaire (QLQ-C38).
Maximal oxygen uptake (VO2max) | On an average 1 week pre surgery
  Cardiopulmonary exercise test
Postoperative complications | Up to five years post surgery
  International Statistical Classification of Diseases and Related Health problems, 10th revision (ICD-10) diagnostic codes, from the patient records
Physical activity level | On an average 1 week pre surgery and three months post surgery
  Activity monitor (SenseWear) to measure level of daily physical activity
In-hospital time | Up to 12 months post surgery
  Number of days in hospital from the patient records

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, PhD, MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Public Health and General Practice, Trondheim, Norway